CLINICAL TRIAL: NCT07250503
Title: Impact of Wearing Two Different Implant Retained Mandibular Overdentures on Occlusal Force Distribution and Denture Retention (Randomized Clinical Trial)
Brief Title: Compare the Difference in Occlusal Force Distribution and Denture Retention Using 2 Different Denture Base Materials in Implant Retained Overdenture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Noha Taha Kamel Taha Alloush, Lecturer, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28.4.24
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Edentulous Alveolar Ridge In Mandible; Complete Edentulism; Dental Implant; Attachments; Implant Retained Overdenture; Edentulous Mouth
Keywords: Completely edentulous patients; Dental Implants; Edentulous Ridge
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandibular complete dentures processed into heat cured acrylic resin (Active Comparator): Mandibular complete dentures made of heat-cured acrylic resin (PMMA). In the mandible, two implants were inserted in the symphyseal area and retained by Equator attachments.
  Interventions: Procedure: Conventional acrylic resin denture
- Mandibular thermoplastic nylon denture (Experimental): Mandibular overdentures were made of the flexible acrylic resin breflex, In the mandible, two implants were inserted in the symphyseal area and retained by Equator attachments.
  Interventions: Procedure: Flexible resin denture

INTERVENTIONS:
Procedure: Conventional acrylic resin denture — Mandibular complete dentures made of heat-cured acrylic resin (PMMA). In the mandible, two implants were inserted in the symphyseal area and retained by Equator attachments.
  Arms: Mandibular complete dentures processed into heat cured acrylic resin
Procedure: Flexible resin denture — Mandibular overdentures were made of the flexible acrylic resin breflex, In the mandible, two implants were inserted in the symphyseal area and retained by Equator attachments
  Arms: Mandibular thermoplastic nylon denture

SUMMARY:
The global increase in the aging population has led to a rise in total edentulism, which remains a major public health concern. two-implant-retained mandibular overdentures have been regarded as the standard of care, offering superior retention, stability, comfort, and masticatory efficiency compared to conventional dentures. Among available attachment systems-bar, ball, stud, and magnet-the Equator attachment has gained popularity due to its low vertical profile, suitability for limited inter-occlusal space, and ease of handling.

Assessment of masticatory performance and occlusal balance can be objectively measured using devices such as bite force analyzers and the computerized T-Scan system, which quantifies occlusion and disocclusion times.

Conventional heat-cured polymethyl methacrylate (PMMA) remains the most widely used denture base material; however, it has mechanical and biological limitations. Flexible denture base materials have been introduced to overcome these drawbacks by enhancing adaptation, distributing occlusal loads more evenly, and improving comfort and retention.

DETAILED DESCRIPTION:
24 Patients will be randomly and equally divided into two treatment groups:

1. Group 1: Each patient in this group will receive conventional maxillary and mandibular complete dentures made of heat-cured acrylic resin PMMA. In the mandible, two implants were inserted in the symphyseal area and retained by equator attachments.
2. Group 2: Patients in this group received the same type of treatment as the patients in group 1, but the mandibular overdentures were made of the flexible acrylic resin "breflex" The present study will be performed to compare the difference in retention, occlusal force distribution, occlusion and disocclusion time, and bite force for implant retained mandibular over denture using PMMA and flexible dentures base materials

ELIGIBILITY:
Inclusion Criteria:

1. All patients age must range from 60-70 years old.
2. All patients' ridges should be covered with firm mucosa free from any signs of inflammation or ulceration and exhibit adequate height and width of the residual alveolar ridge.
3. Patients should be free from any metabolic or bone disorder that contraindicate implant installation.
4. All patients must have sufficient inter arch space

Exclusion Criteria:

1. Patients with oral or systemic diseases.
2. Patients with xerostomia or excessive salivation.
3. Patients with parafunctional habits (bruxism or clenching).
4. Heavy smoker or alcoholic patients.
5. Patients with history of temporo-mandibular dysfunction.
6. Patients with brain disorders or psychiatric disorders

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Occlusal force distribution | Follow up visits were scheduled at denture insertion, 6, and 12 months
  Occlusal force distribution will be measured by T-Scan, The latest version (T-Scan III) provides a dynamic visual evaluation of a patient's occlusion from initial tooth contact to maximum intercuspation. The system records relative force values and allows objective quantitative evaluation of occlusal balance by recording numerical values for occlusion and disocclusion times

SECONDARY OUTCOMES:
Retention of lower denture | Follow up visits were scheduled at denture insertion, 6, and 12 months
  Retention of lower denture will be measured using digital force gauge, Retention will be measured using digital force gauge A digital force meter was used to measure denture resistance to vertical displacement (i.e., retention) by applying a pulling force on a metal hook located in the geometric center of each mandibular conventional denture that was identified on the lower cast at the intersection of three lines bisecting the angles of the triangle, formed by both retromolar pads and the midline. Measurement of mandibular denture retention: The patient was instructed to place his head on chin rest and occlusal plane was set parallel to the floor. Tongue freedom was checked then and three minutes seating time was allowed before taking the measurements. A vertical pulling force was applied using the metallic probe of the digital force-meter that was attached to the hook present at the geometric center of mandibular denture. Average value of six readings was recorded.
occlusion time | Follow up visits were scheduled at denture insertion, 6, and 12 months
  occlusion and disocclusion time will be measured by T-Scan, The latest version (T-Scan III) provides a dynamic visual evaluation of a patient's occlusion from initial tooth contact to maximum intercuspation. The system records relative force values and allows objective quantitative evaluation of occlusal balance by recording numerical values for occlusion times
Biting force | Follow up visits were scheduled at denture insertion, 6, and 12 months
  Biting force will be measured by bite force meter
Disocclusion time | Follow up visits were scheduled at denture insertion, 6, and 12 months
  will be measured by T-Scan, The latest version (T-Scan III) provides a dynamic visual evaluation of a patient's occlusion from initial tooth contact to maximum intercuspation. The system records relative force values and allows objective quantitative evaluation of occlusal balance by recording numerical values for disocclusion times

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol and Clinical Study Report
Supporting Information: Study Protocol, CSR
Time Frame: Start Date: After publication End Date: 3 years
Access Criteria: After publication through the corresponding author